CLINICAL TRIAL: NCT02481557
Title: Effects of an Oxalate Containing Product on Dentinal Hypersensitivity With Dental Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015069
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

ARMS (2):
- Oxalate Salt Solution (Experimental): Professionally applied
  Interventions: Device: Oxalate Salt Solution
- No Treatment (No Intervention): No Treatment

INTERVENTIONS:
Device: Oxalate Salt Solution — Applied by dentist
  Arms: Oxalate Salt Solution

SUMMARY:
This study will assess sensitivity during a dental prophylaxis with or without the use of a potassium oxalate salt solution.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* sign an informed consent form and be given a copy
* be in good general health as determined by the Investigator/designee
* agree to delay any elective dentistry, and to report any dentistry received during the course of the study
* agree to not participate in any other oral care study for the duration of this study
* agree to return for scheduled visits and follow all study procedures
* have at least one tooth with a Schiff sensitivity score of at least 1 in response to air challenge and a Yeaple Probe score of 10-40 in response to tactile challenge.

Exclusion Criteria:

* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession
* active treatment for periodontitis
* any diseases or conditions that might interfere with the subject safely completing the study
* inability to undergo study procedures
* fixed orthodontic appliances

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstone Research Group, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Treatment: No study treatment
Period: Overall Study
Arm/Group | Oxalate Salt Solution | No Treatment
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxalate Salt Solution | No Treatment | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (14.14) | 34.5 (10.11) | 34.5 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 4 | 2 | 6
  Ethnicity: Asian Oriental | 4 | 2 | 6
  Ethnicity: Black | 1 | 4 | 5
  Ethnicity: Caucasian | 6 | 8 | 14
  Ethnicity: Multi-Racial | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Air Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A negative change from Baseline score represents a decrease in sensitivity from baseline. The mean change from Baseline was calculated for this measure.
Time Frame: 10 Minutes
Population: Thirty-Six (36) subjects received products. Thirty-Six (36) subjects completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxalate Salt Solution | No Treatment
Number analyzed (Participants) | 17 | 19
Units on a scale | -0.412 (0.537) | -0.132 (0.403)

2. Secondary Outcome: Change From Baseline for Yeaple Probe
Description: Tactile Threshold was measured using a Yeaple probe. Testing was performed beginning at 10 g. The examiner recorded tactile scores for responding teeth. After treatment, testing began at 10 g and increase by 10 g to a maximum of 50 g. The higher the tactile threshold, the less sensitive the tooth. Each successive challenge increased until a "yes" response was repeated. If a second "yes" was not obtained, the force setting was increased to the next step and continued until a force was found which elicited two consecutive "yes" responses and was recorded as the threshold on the Tactile Sensitivity Score form. The mean change from Baseline was calculated for this measure.
Time Frame: 10 Minutes
Population: Thirty-six (36) subjects received study products. Thirty-six (36) subjects completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxalate Salt Solution | No Treatment
Number analyzed (Participants) | 17 | 19
Units on a scale | 10.000 (8.101) | 1.316 (6.634)

ADVERSE EVENTS:
Arm/Group | Oxalate Salt Solution | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes